CLINICAL TRIAL: NCT05952076
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of Bi-26 (Strain of Bifidobacterium Longum, B. Infantis) Supplementation Versus Placebo on Weight Gain in Underweight Infants
Brief Title: Impact of Bi-26 Supplementation on Weight Gain in Underweight Infants
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Gates Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Gates MRI-MNK01-301
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Underweight; Paediatrics
Keywords: Weight-for-age Z score; Underweight infants; Bifidobacterium longum, B. infantis; Bi-26 supplementation
MeSH Terms: conditions — Thinness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bi-26 supplementation (Experimental): Bi-26 administered daily.
  Interventions: Dietary Supplement: B. infantis Bi-26
- Placebo (Placebo Comparator): Maltodextrin: Placebo administered daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: B. infantis Bi-26 — A once-daily oral dose of Bi-26 will be provided to infants for 28 days.
  Arms: Bi-26 supplementation
Dietary Supplement: Placebo — A once-daily oral dose of placebo maltodextrin will be provided to infants for 28 days
  Arms: Placebo

SUMMARY:
The burden of disease experienced by underweight children is significant, particularly in low- and middle-income countries. Gut dysbiosis, an imbalance in microbial composition, is thought to play a role in nutrient malabsorption leading to underweight infants and failure to thrive. Bifidobacterium longum subspecies infantis (B. infantis) is a commensal bacterial strain important in the breakdown of human milk oligosaccharides (HMOs). A decrease in abundance or absence of B. infantis could lead to inadequate HMO processing, elevating intestinal pH and increasing the risk of pathogen overgrowth. Bi-26 is a B. infantis probiotic strain that is being evaluated in this study for its impact on weight gain and other health outcomes in underweight infants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be between 30 days and 120 days of age (inclusive), at the time of enrollment (study Day 1)
* Hospitalized for acute non-surgical illness
* Completed acute stabilization phase of treatment, including fluid rehydration and antibiotic course, prior to enrollment (study Day 1)
* WAZ at enrollment (study Day 1) is less than negative 2 (<-2)
* Any sex
* Participant's parent(s)/legal guardian is capable of giving informed consent which includes agreement to comply with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol
* Participant's parent(s)/legal guardian agrees to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and have no current plans to relocate from the study area for the duration of the study
* Participant's parent(s)/legal guardian has easy access to reliable refrigeration (for storage of investigational product)
* Participant receives some feedings from breastmilk and mother intends to continue breastfeeding.

Exclusion Criteria:

* Congenital condition (suspected or confirmed) that the investigator considers likely to interfere with feeding or with normal growth and development
* Infant has not been discharged from hospital since birth or has not been at home for at least one week since birth
* Infant hospitalized with septic shock during current hospitalization
* Infant required mechanical ventilation during current hospitalization
* Infant with acute kidney injury on hospital admission
* Infant with severe jaundice and suspected kernicterus
* Infant receiving treatment for suspected or confirmed tuberculosis, or suspected or confirmed human immunodeficiency virus (HIV) infection
* Ongoing infant antibiotic (e.g. as prophylaxis in sickle cell disease) and/or probiotic usage
* Ongoing maternal antibiotic and/or probiotic usage for breast-feeding infants
* Inability of participant's parent(s)/legal guardian to comply with protocol requirements, as per investigator assessment.

Ages: 30 Days to 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2024-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gates MRI, Study Director — Gates Medical Research Institute
Locations (5):
- Pakistan (5):
  - Medical Facility A, Islamabad, Islamabad
  - Medical Facility B, Islamabad, Islamabad
  - Medical Facility C, Islamabad, Islamabad
  - Medical Facility, Lahore, Punjab Province
  - Medical Facility, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: Yes
All IPD data that underlie results in a publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: This will be done within 12months of the study completion date.
Access Criteria: Anonymized participant level data may be shared with external researchers in accordance with the trial participants' written and executed informed consent document and any local or applicable regulations on data sharing. Qualified researchers may submit a request for anonymized participant level data along with a research proposal to Gates MRI for review. The types of supporting information that could be shared with external researchers include: the Study Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report, and analytic code. A data sharing agreement must be in place before any clinical trial data are shared. There are additional circumstances that may prevent the sharing of data with external researchers, including but not limited to contractual obligations to existing partners and any restrictions imposed by regulatory bodies.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 3, randomized, double-blind study that evaluated the impact of Bi-26 (strain of Bifidobacterium longum, B. infantis) supplementation on weight gain in underweight infants.
Pre-assignment Details: A total of 40 participants were enrolled from 1 country and were randomized 1:1 in experimental and placebo groups.
Groups:
- Bi-26 Supplementation: Participants received Bi-26 supplementation once-daily orally for 28 days.
- Placebo: Participants received placebo (maltodextrin) once-daily orally for 28 days.
Period: Overall Study
Arm/Group | Bi-26 Supplementation | Placebo
Started | 20 | 20
Completed | 19 | 18
Not Completed | 1 | 2
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population comprised of all participants randomly assigned to study intervention, who received any dose, including a partial dose, of the study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bi-26 Supplementation | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Days] | 57.6 (21.1) | 66.6 (23.6) | 62.1 (22.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 20 | 20 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weight-for-age Z Score (WAZ) at Day 56
Description: The Weight-for-Age Z-score (WAZ) is an anthropometric measure used to classify a child's nutritional status. The WAZ measures the number of standard deviations of a child's actual weight from the median weight of children of the same age based on the World Health Organization (WHO) child growth standards (reference population). WAZ of 0 represents the median weight for age in the reference population. WAZ ≥-3 to <-2 standard deviations below the WHO child growth standards median is considered moderately underweight and WAZ <-3 is considered severely underweight. Least Squares Mean, 95% Confidence Interval, and p-value was derived from mixed model repeated measures with treatment and visit as factors and baseline WAZ, baseline age (days), and study intervention compliance as covariates. The treatment*visit interaction terms were included and used to estimate the adjusted mean difference in Change from Baseline in WAZ between Bi-26 and Placebo.
Time Frame: Baseline (Day 1) to Day 56
Population: Modified Intention to Treat Population comprised of all participants randomly assigned to study intervention, who received any dose, including a partial dose of the study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Bi-26 Supplementation | Placebo
Number analyzed (Participants) | 20 | 20
Z-score | 0.78 [0.39 to 1.17] | 0.67 [0.28 to 1.06]
Statistical Analysis 1: Comparison: Bi-26 Supplementation vs Placebo; Test type: Other; p = 0.6863, Mixed Models Analysis; See Estimation Comments; Adjusted mean difference = 0.11, 95% CI 2-sided [-0.44 to 0.67] — The mixed model included treatment and visit as factors, including the interaction term, and was adjusted by baseline WAZ and baseline age (days). A random intercept for participant was included

2. Secondary Outcome: Change From Baseline in Weight to Day 56
Description: Weight (grams) was summarized using descriptive statistics. Baseline (Day 1) was defined as the last available value prior to the participant receiving the first dose of the study intervention. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) to Day 56
Population: Modified Intention to Treat Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Grams
Arm/Group | Bi-26 Supplementation | Placebo
Number analyzed (Participants) | 20 | 20
Grams | 1491.47 [1233.45 to 1749.48] | 1382.17 [1123.95 to 1640.39]
Statistical Analysis 1: Comparison: Bi-26 Supplementation vs Placebo; Test type: Other; p = 0.5567, Mixed Models Analysis; See Estimation Comments; Adjusted mean difference = 109.30, 95% CI 2-sided [-259.76 to 478.36] — The mixed model included treatment and visit as factors, including the interaction term, and was adjusted by baseline weight (grams) and baseline age (days). A random intercept for participant was included

3. Secondary Outcome: Change From Baseline in WAZ Over Time Through Day 90
Description: as for outcome 1
Time Frame: Baseline (Day 1) to Day 90
Population: Modified Intention to Treat Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Bi-26 Supplementation | Placebo
Number analyzed (Participants) | 20 | 20
Z-score | 1.09 [0.70 to 1.48] | 1.00 [0.60 to 1.39]
Statistical Analysis 1: Comparison: Bi-26 Supplementation vs Placebo; Test type: Other; p = 0.7275, Mixed Models Analysis; See Estimation Comments; Adjusted mean difference = 0.10, 95% CI 2-sided [-0.46 to 0.66] — The mixed model included treatment and visit as factors, including the interaction term, and was adjusted by baseline WAZ, baseline age (days) and study intervention compliance. A random intercept for participant was included

4. Secondary Outcome: Percentage of Participants With a ≥ 0.3, ≥ 0.4, and ≥ 0.5 Change in WAZ From Baseline at Day 56
Description: The Weight-for-Age Z-score (WAZ) is an anthropometric measure used to classify a child's nutritional status. The WAZ measures the number of standard deviations of a child's actual weight from the median weight of children of the same age based on the World Health Organization (WHO) child growth standards (reference population). WAZ of 0 represents the median weight for age in the reference population. WAZ ≥-3 to <-2 standard deviations below the WHO child growth standards median is considered moderately underweight and WAZ <-3 is considered severely underweight.
Time Frame: Baseline (Day 1) to Day 56
Population: Per-Protocol (PP) Population comprised of all participants randomly assigned to study intervention, who received the study intervention, have a Day 90 visit, and did not substantially deviate from the protocol procedures.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bi-26 Supplementation | Placebo
Number analyzed (Participants) | 16 | 14
Percentage of participants
  Increase of >= 0.3 units | 87.5 [64.5 to 97.8] | 64.3 [37.6 to 85.6]
  Increase of >= 0.4 units | 87.5 [64.5 to 97.8] | 64.3 [37.6 to 85.6]
  Increase of >= 0.5 units | 68.8 [43.7 to 87.5] | 64.3 [37.6 to 85.6]

5. Secondary Outcome: Percentage of Participants Who Achieved a Score of WAZ > -2 at Day 56
Description: as for outcome 4
Time Frame: At Day 56
Population: PP Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bi-26 Supplementation | Placebo
Number analyzed (Participants) | 16 | 14
Percentage of participants | 19 [5.0 to 43] | 14 [2.5 to 39.7]

6. Secondary Outcome: Percentage of Participants Re-hospitalized
Description: Hospitalizations are due to acute non-surgical illness. Percentage of participants re-hospitalized at Day 56 has been presented
Time Frame: Baseline to Day 56
Population: Safety Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bi-26 Supplementation | Placebo
Number analyzed (Participants) | 20 | 20
Percentage of participants | NA [NA to NA] — Data was not available as there were no events reported in Bi-26 supplementation arm that resulted in re-hospitalization. | 20 [5.7 to 43.7]

7. Secondary Outcome: Number of Participants Reporting Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE is considered treatment emergent if it started on or after the date of first dose of study intervention administration. Serious TEAE is any untoward medical occurrences at any dose of study medication that: results in death; is life threatening; requires inpatient hospitalization or causes prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect and is an important medical event.
Time Frame: Up to Day 90
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Bi-26 Supplementation | Placebo
Number analyzed (Participants) | 20 | 20
Participants
  Any TEAE | 8 | 16
  Any serious TEAE | 1 | 5

8. Secondary Outcome: Percentage of Participants With Presence of B. Infantis in Stool
Description: Stool samples were collected at defined time points to analyze the present of B.infantis.
Time Frame: At Days 1, 28, 56 and 90
Population: PP Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bi-26 Supplementation | Placebo
Number analyzed (Participants) | 16 | 14
Percentage of participants
  Day 1 | 62.5 [37.6 to 83.2] | 50.0 [25.1 to 74.9]
  Day 28 | 100.0 [82.9 to 100.0] | 57.1 [31.1 to 80.4]
  Day 56 | 100.0 [82.9 to 100.0] | 57.1 [31.1 to 80.4]
  Day 90 | 93.8 [72.8 to 99.7] | 57.1 [31.1 to 80.4]

ADVERSE EVENTS:
Time Frame: Up to 90 Days
Description: TEAEs and serious AEs were collected in Safety Population.
Arm/Group | Bi-26 Supplementation | Placebo
All-Cause Mortality (participants affected / at risk) | 1/20 | 1/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 5/20
Other Adverse Events (participants affected / at risk) | 7/20 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bi-26 Supplementation (N=20) | Placebo (N=20)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Pneumonia measles (Infections and infestations) | 0 | 1
Death (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bi-26 Supplementation (N=20) | Placebo (N=20)
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 4 | 8
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Pyrexia (General disorders) | 0 | 3
Nasopharyngitis (Infections and infestations) | 1 | 2
Acarodermatitis (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 1
Conjunctivitis viral (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Measles (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT05952076/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT05952076/SAP_001.pdf